CLINICAL TRIAL: NCT01613170
Title: A Combined Treatment Program for the Symptoms of Urinary Urgency and Frequency With Toviaz and Premarin Vaginal Cream
Brief Title: Premarin Versus Toviaz for Treatment of Overactive Bladder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cleveland Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, G. Willy Davila, Chairmain of Department of Gynecology and Head of Section of Urogynecology, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11074
Record Dates: First submitted 2012-05-24; First posted 2012-06-07 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Vaginal Estrogen; Anticholinergics; Antimuscarinics
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine; Estrogens, Conjugated (USP); Estrogens

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Toviaz and Premarin Vaginal Cream (Experimental): Toviaz 4 mg PO q day and premarin cream 1 g per vagina 2 times a week.
  Interventions: Drug: Toviaz; Drug: Premarin
- Toviaz , Placebo Premarin Vaginal Cream (Placebo Comparator): Toviaz 4 mg PO q day and placebo cream 1 g per vagina 2 times a week.
  Interventions: Drug: Toviaz; Drug: Placebo cream

INTERVENTIONS:
Drug: Toviaz — Toviaz 4mg daily
  Other Names: fesoteridine
Drug: Premarin — Premarin cream 1 g per vagina twice weekly
  Other Names: estrogen, conjugated vaginal
  Arms: Toviaz and Premarin Vaginal Cream
Drug: Placebo cream — Placebo cream 1 g per vagina twice weekly, to mimic Premarin cream
  Other Names: Verba base cream
  Arms: Toviaz , Placebo Premarin Vaginal Cream

SUMMARY:
The use of vaginal estrogen cream in conjunction with Toviaz will be more effective than the use of Toviaz alone for the treatment of overactive bladder.

DETAILED DESCRIPTION:
Participants will be randomized to two treatment arms with 45 patients enrolled in each study arm: Toviaz and Premarin Vaginal Cream and Toviaz and Placebo Premarin Vaginal Cream. The Toviaz will be dosed at 4mg tablet given as a once daily dose. Premarin vaginal cream will be dosed at 1 gram per vagina twice weekly. Compliance will be assessed at the 4-week mark and again at completion of the study, 8 weeks after the commencement of treatment.

The questionnaires chosen for this study have been designed and validated as effective tools to assess and evaluate OAB. Patients will be asked to complete three symptoms questionnaires and a 3-day voiding dairy. The questionnaires include Overactive Bladder Questionnaire (OAB-q), The Patient Perception of Bladder Condition, and Urgency Severity and Impact Questionnaire. The voiding diary and questionnaires will be filled out and collected at the initial visit and again at the end of the study which is defined as 8 weeks after the commencement of treatment.

Additionally, patients will be asked to rate their symptoms associated with urogenital atrophy at the start of the study and then again at 8 weeks. The severity of each symptom will be graded based on a four-point scale (0=none, 1=mild, 2= moderate, 3=severe) and a composite score will then be generated. Examiners will also rate the severity of signs of urogenital atrophy at the first visit and at the conclusion of the study.

An objective evaluation of the effectiveness of the estrogen cream treatment will be accomplished by a pathological evaluation of the vaginal cell samples at the beginning of treatment and then again at the 8 week point. These cells will be collected and analyzed by an independent pathologist to determine the percentage of parabasal, intermediate, and superficial cells and to document the change in these three categories of cells as a result of the vaginal estrogen treatment. A 3-Day voiding diary will be used to document changes from baseline for urinary urgency, frequency, and incontinence episodes. Based on previous studies we predict there will be a 45% improvement on urinary frequency from baseline when using both Toviaz and vaginal Premarin cream. Secondary outcomes will be measured using the following validated questionnaires given at the start of the study and again at completion: OAB-q, Patient Perception of Bladder Condition, Urgency Severity and Impact Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Women defined as at least 12 months since last menstrual period
* OAB symptoms for 6 months or longer with complaints of frequency (8 or more voids in a 24 hour period), and either 6 or more urgency episodes in 24 hours, and either 3 or more urge urinary incontinence episodes per 24 hours.

Exclusion Criteria:

* Current or recent treatment (within the last 6 months) with estrogens
* Past or present history of estrogen dependent neoplasm
* Undiagnosed genital tract bleeding
* Current urinary or vaginal infection
* History of thromboembolic disorders associated with estrogen use
* Commencement or alteration of diuretic therapy within three months of study enrollment
* No contraindications for anticholinergic medical therapy
* No contraindications to estrogen therapy
* Symptoms must not have commenced more than three years prior to menopause
* Post Void Residual must be under or equal to 150 ml
* Recurrent Urinary Tract Infections (3 culture proven UTI's within the past 12 months)
* Not on any other anticholinergic medications for the last 4 weeks
* Painful Bladder Syndrome
* Chronic Pelvic Pain
* Vaginal Prolapse POPQ > stage 2/ maximal prolapse point greater than +1 cm

Ages: 30 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Urinary frequency as measured by a 3 day voiding diary | 1 year
  number of voids per day

SECONDARY OUTCOMES:
Lifestyle Impact of Overactive Bladder as measured using 3 validated questionnaires: OAB-Q, PPBC, and Urgency Severity and Impact Questionnaire | 1 year
  quality of life assessment via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hurtado, MD, Principal Investigator — Cleveland Clinic Florida; Alexandriah Alas, MD, Study Director — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No